CLINICAL TRIAL: NCT04791228
Title: A Pilot Study of Lyso-thermosensitive Liposomal Doxorubicin (LTLD, ThermoDox®) and Magnetic Resonance-Guided High Intensity Focused Ultrasound (MR-HIFU) for Treatment of Relapsed or Refractory Solid Tumors
Brief Title: A Pilot Study of Thermodox and MR-HIFU for Treatment of Relapsed Solid Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment.
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, AeRang Kim, Oncologist, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU Thermodox PII
Record Dates: First submitted 2021-02-22; First posted 2021-03-10 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumors; Soft Tissue Sarcoma; Ewing Sarcoma; Malignant Epithelial Neoplasm; Rhabdomyosarcoma; Wilms Tumor; Hepatic Tumor; Germ Cell Tumor; Bone Metastases
Keywords: Relapsed/refractory solid tumors; High Intensity Focused Ultrasound; Lyso-thermosensitive Liposomal Doxorubicin; ThermoDox
MeSH Terms: conditions — Sarcoma; Sarcoma, Ewing; Carcinoma; Rhabdomyosarcoma; Wilms Tumor; Carcinoma, Hepatocellular; Neoplasms, Germ Cell and Embryonal; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- All Patients (Experimental): LTLD 50 mg/m2 will be administered intravenously over 30 minutes on day 1 of every 21-day cycle. MR-HIFU hyperthermia will follow infusion (+/- 30 minutes) for one hour to a target area with a target temperature of 40-45°C followed by ablation therapy (>55°C). The HIFU hyperthermia regimen will have a duration of at least 60 minutes and will then be followed by ablation therapy. Patients may receive up to a total of 6 cycles. Subsequent treatment cycles may treat alternative target lesions. Disease status will be evaluated using standard imaging techniques (CT/MR) post each cycle.
  Interventions: Device: Magnetic Resonance-Guided High Intensity Focused Ultrasound; Drug: Lyso-thermosensitive Liposomal Doxorubicin

INTERVENTIONS:
Device: Magnetic Resonance-Guided High Intensity Focused Ultrasound — Magnetic resonance (MR)-guided high intensity focused ultrasound (HIFU) provides precise and controlled delivery of heat by focusing ultrasound energy inside a lesion using an external applicator without the need for a scalpel or needle.
  Additional therapeutic advantages of this modality include its range of bioeffects, including both high temperature tumor ablation via coagulative necrosis, and effects of lower temperature, mild hyperthermia that can help to enhance local drug delivery to tumors. Both tumor ablation and hyperthermia may be employed to potentiate the effects of chemotherapy.
  Other Names: MR-HIFU
Drug: Lyso-thermosensitive Liposomal Doxorubicin — LTLD combines doxorubicin with lyso-thermosensitive liposomes that can selectively deliver drug to tumors and when exposed to temperatures greater than 40°C, rapidly and locally releases doxorubicin in high concentrations from systemically administered LTLD.
  If combined with hyperthermia, doxorubicin will be released in the heated tumor margins and in any areas within the tumor that were not completely ablated and increase the likelihood of complete tumor necrosis. LTLD will extend tumor cell death to the hyperthermic regions in the peri-ablation zones and minimize the possibility of incomplete ablation or tumor recurrence.
  Other Names: LTLD; ThermoDox

SUMMARY:
This is a pilot study of LTLD with MR-HIFU hyperthermia followed by ablation in subjects with refractory/relapsed solid tumors.

DETAILED DESCRIPTION:
LTLD is a heat-activated formulation of liposomal doxorubicin that releases the drug when exposed to hyperthermic conditions (40-45°C). This novel agent has been well tolerated in adults with similar toxicity profile to doxorubicin. MR-HIFU offers a non-invasive and non-ionizing ability to selectively heat large tissue volumes. Thus, MR-HIFU is a promising technology for triggering doxorubicin release from LTLD. The investigator's approach involves continuous maintenance of the target at mild hyperthermia with MR-HIFU following LTLD infusion. Following hyperthermia, the investigators will deliver ablation therapy (>55°C) to targeted areas of tumor where feasible and safe. Addition of this ablation therapy after mild-hyperthermia-triggered drug delivery with LTLD has the potential to significantly potentiate chemotherapy with minimal additional adverse effects to improve local control and drug delivery without increasing toxicity.

ELIGIBILITY:
Inclusion Criteria:

* AGE: ≥ 12 years of age.
* DIAGNOSIS: Histologically confirmed malignant solid tumors
* TUMOR LOCATION: Patient must have at least one tumor located in areas accessible to HIFU, which will be defined as the target lesion(s). Target lesions must be reachable within the normal safety margins of HIFU as specified in the instructions for use.
* TARGET LESION(S): Radiographically measurable/evaluable solid tumor target lesion(s).
* THERAPEUTIC OPTIONS:

  - Malignant Tumor: The patient's cancer must have relapsed after or failed to respond to frontline curative therapy and there must not be other potentially curative treatment options available.
* PRIOR THERAPY:

  * Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering on this study.
  * No limitation on the number of prior chemotherapy regimens that the patient may have received prior to study entry.
  * Myelosuppressive chemotherapy: The last dose of all myelosuppressive anticancer drugs must be at least 3 weeks prior to study entry (6 weeks for prior nitrosoureas) Prior treatment with anthracyclines is allowed as long as total cumulative dose is ≤ 450 mg/m2.
  * Immunotherapy: The last dose of immunotherapy (monoclonal antibody or vaccine) must be at least 3 weeks prior to study entry.
  * Biologic (anti-cancer agent): The last dose of all biologic agents for the treatment of the patient's cancer (such as retinoids or tyrosine kinase inhibitors) must be at least 7 days prior to study entry.
  * Radiation therapy: The last dose of radiation to more than 25% of marrow containing bones (pelvis, spine, skull) must be at least 4 weeks prior to study entry. The last dose of all other local palliative (limited port) radiation must be at least 2 weeks prior to study entry.
  * Stem Cell Transplantation. At least 42 days post-autologous stem cell transplant or at least 90 post-allogeneic transplant and recovered from toxicities without evidence of graft versus host disease and on stable doses of immunosuppressive medications if required.
  * Growth Factors. The last dose of colony stimulating factors, such as filgrastim, sargramostim, and erythropoietin, must be at least 1 week prior to study entry, the last dose of long-acting colony stimulating factors, such as pegfilgrastim, must be at least 2 weeks prior to study entry.
* CONCURRENT THERAPIES:

  - No other anti-cancer therapy (chemotherapy, biological therapy, radiation therapy) is permitted.
* PERFORMANCE STATUS:

  * Lansky/Karnofsky performance level ≥ 50% (See Appendix I).
  * Patients who are unable to walk because of paralysis or motor weakness, but who are up in a wheelchair will be considered ambulatory for the purpose of calculating the performance score.
* HEMATOLOGIC FUNCTION:

  * Peripheral absolute neutrophil count (ANC) of ≥ 1000/µL.
  * Platelet count ≥ 75,000/µL (transfusion independent (no transfusion within at least 7 days prior to enrollment)).
* HEPATIC FUNCTION:

  * Total bilirubin must be ≤ 1.5 times the upper limit of normal (ULN) for age and gender.
  * SGPT (ALT) must be ≤ 3.0 times the upper limit of normal for age.
* RENAL FUNCTION: Serum creatinine ≤ ULN for age/sex OR a creatinine clearance ≥60 mL/min/1.73 m2.
* CARDIAC FUNCTION: Adequate Cardiac Function with Ejection Fraction > 50% by echocardiogram.

Exclusion Criteria:

* Clinically significant unrelated systemic illness, such as serious infections, hepatic, renal or other organ dysfunction, which in the judgment of the Principal or Associate Investigator would compromise the patient's ability to tolerate study interventions.
* Patients who are pregnant or breast-feeding are not eligible for this study due to risks of fetal and teratogenic adverse events seen in animal/human studies with doxorubicin. Negative pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method beginning at the signing of informed consent and until at least 30 days after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or designated associate.
* Implant or prosthesis within the path of the HIFU beam.
* Target pathway <1 cm from nerve plexus, spinal canal, or bowel.
* Target lesion in the skull.
* Inability to undergo MRI and/or contraindication for MRI.
* Inability to tolerate stationary position during HIFU.
* Previous history of hypersensitivity to doxorubicin or its liposomal formulations.
* Patients currently receiving other anticancer agents.
* Patients currently receiving other investigational agents.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Primary objective 1: Response of treated target lesion(s) assessed by CT or MRI | At the end of every 21-day cycle
  The Response Evaluation Criteria in Solid Tumors (RECIST v1.1) will be used
Primary objective 2: The number of participants with treatment-related adverse events as assessed by the Common Terminology Criteria of Adverse Events (CTCAE) v.5 | Up to thirty days after last dose of protocol therapy
  CTCAE v.5 will be used

OTHER OUTCOMES:
Exploratory objective 1: Response of non-target lesion(s) assessed by CT or MRI | At the end of every 21-day cycle
  Lesions that are evaluable or measurable but not in the treated location(s) will be collected
Exploratory objective 2: Participant reported target tumor pain intensity assessed using the Numerical Rating Scale-11 (NRS-11) | At the end of every 21-day cycle
  The NRS-11 consists of a 11-point numeric scale to assess pain intensity from 0 (no pain) to 10 (worst pain)
Exploratory objective 3: Participant reported impact of pain on daily activities assessed using the PROMIS Pain Interference Scale (PROMIS-PI) | At the end of every 21-day cycle
  The PROMIS-PI consists of 8 questions on pain. Each question will be rated from 0 (never), 1 (almost never), 2 (sometimes), 3 (often), and 4 (almost always)
Exploratory objective 4: Blood samples taken to see adaptive immune response and immune suppression | At 1 day and 1 week after MR-HIFU treatment on first 21-day cycle
  To determine changes in pharmacodynamics of immune markers

CONTACTS AND LOCATIONS:
Overall Officials: AeRang Kim, MD, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States